CLINICAL TRIAL: NCT02503189
Title: A Phase III Study of KCT-0809 in Dry Eye Patients With Sjögren's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KCT1301
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Dry Eye With Sjögren's Syndrome
Keywords: Dry eye syndromes; Corneal diseases; Conjunctival diseases
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases; Conjunctival Diseases

ARMS (2):
- KCT-0809 (Experimental)
  Interventions: Drug: KCT-0809 ophthalmic solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KCT-0809 ophthalmic solution
  Arms: KCT-0809
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the superiority of KCT-0809 to placebo, and to evaluate safety in dry eye patients with Sjögren's syndrome

ELIGIBILITY:
Inclusion Criteria:

* Dry eye patients with Sjögren's syndrome
* Corneal and conjunctival damage

Exclusion Criteria:

* Severe ophthalmic disorder
* Punctal plugs or surgery for occlusion of the lacrimal puncta

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Score of the corneal staining | 12 weeks

SECONDARY OUTCOMES:
Score of the conjunctival staining | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo and Other Japanese City, Japan